CLINICAL TRIAL: NCT05941026
Title: Developing Nursing Students' Intercultural Sensitivity Levels: A Randomized Controlled Experimental Study
Brief Title: Developing Nursing Students' Intercultural Sensitivity Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, ÖNER ALTINTOP, Master (PhD Student), Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Intercultural Sensitivity
Record Dates: First submitted 2023-06-21; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Nursing Caries; Education
Keywords: Nursing; Student; Culture; Intercultural; Sensitivity; Education
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Following recruitment, students were divided into a study and a control group by randomization (1:1 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arms (Experimental): Nursing students who were in the experimental group during the application phase of the study were given training to develop their intercultural sensitivity levels based on Leninger's Intercultural Nursing Theory. Data were collected at the beginning of the four-week online training, at the end of the training, and one month after the training.
  Interventions: Other: Structured education
- Control groups (No Intervention): No application was made to the control group within the scope of the research. Data were collected simultaneously with only the experimental group.

INTERVENTIONS:
Other: Structured education — The educational content of the research was created by the researcher in line with the literature and expert opinions and covers the following topics.
  Educational subjects
  1. Culture and Concepts Related to Culture
  2. Culture/Cultural Characteristics and Cultural Elements in Terms of Social Structure
  3. Cultural Factors Affecting Health and Disease
  4. Concepts and Practices Related to the Field of Study
  The training is an online training and continued via video conference, and a session invitation was sent to the participants before each session. In addition, after the training, brochures containing the training topics of each week were prepared and delivered to the participants. The trainings were conducted by the researcher in a total of four sessions (each session 20 minutes) once a week during the training process. During the training, the questions of the participants were answered.
  Arms: Arms

SUMMARY:
This study; This is a randomized controlled experimental type study designed to improve the intercultural sensitivity levels of nursing students.

DETAILED DESCRIPTION:
Cultural sensitivity is extremely important for healthcare professionals. Understanding cultural differences can help build a trusting relationship between patients and healthcare professionals. This increases patient satisfaction and improves the quality of health services.

This work; This is a randomized controlled experimental type study designed to improve the intercultural sensitivity levels of nursing students.

Intercultural sensitivity training does not affect the intercultural sensitivity level of nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Being a student of Aydın Adnan Menderes University Nursing Department
* Having successfully completed the basic practical courses of the first three classes
* Being enrolled in one of the Public Health Nursing or Mental Health and Diseases Nursing courses from the fourth year
* Volunteer to participate in the study

Exclusion Criteria:

• Not completing the training sessions of the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Intercultural Sensitivity Scale and Personel Questions | Pre-test (Before the training)
  The scale was developed by Chen and Starosta and was adapted to Turkish in 2010. It consists of twenty-four items and includes five emotional dimensions necessary to measure intercultural sensitivity. The scale has five dimensions: responsibility in communication, respect for cultural differences, self-confidence in communication, enjoying communication, and being careful in communication. The scale has a 5-point Likert-type rating. As the score obtained from the scale increases, the level of sensitivity increases. The Cronbach's alpha value of the scale was determined as 0.90.
Intercultural Sensitivity Scale | four weeks after the pre-test (at the end of the training)
  The scale was developed by Chen and Starosta and was adapted to Turkish in 2010. It consists of twenty-four items and includes five emotional dimensions necessary to measure intercultural sensitivity. The scale has five dimensions: responsibility in communication, respect for cultural differences, self-confidence in communication, enjoying communication, and being careful in communication. The scale has a 5-point Likert-type rating. As the score obtained from the scale increases, the level of sensitivity increases. The Cronbach's alpha value of the scale was determined as 0.90.
Intercultural Sensitivity Scale | eight weeks after the pre-test (and one month after the training)
  The scale was developed by Chen and Starosta and was adapted to Turkish in 2010. It consists of twenty-four items and includes five emotional dimensions necessary to measure intercultural sensitivity. The scale has five dimensions: responsibility in communication, respect for cultural differences, self-confidence in communication, enjoying communication, and being careful in communication. The scale has a 5-point Likert-type rating. As the score obtained from the scale increases, the level of sensitivity increases. The Cronbach's alpha value of the scale was determined as 0.90.

CONTACTS AND LOCATIONS:
Overall Officials: Öner ALTINTOP, MsC, Study Chair — Aydın Adnan Menderes University Institute of Health Sciences Department of Public Health Nursing
Locations (1):
- Aydın Adnan Menderes University Institute of Health Sciences Department of Public Health Nursing, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.